CLINICAL TRIAL: NCT04920695
Title: The Impact of Inhaled Nitric Oxide (iNO) on the Neurophysiological Mechanisms of Dyspnea in Chronic Thromboembolic Disease and Post-Pulmonary Embolism (Post-PE) Related Dyspnea
Brief Title: Inhaled Nitric Oxide (iNO) in Post-Pulmonary Embolism (Post-PE)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Denis O'Donnell (Other)
Responsible Party: Sponsor-Investigator, Dr. Denis O'Donnell, Doctor, Professor, Director of RIU, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: DMED 2415-20
Record Dates: First submitted 2021-01-21; First posted 2021-06-10 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Dyspnea; Pulmonary Embolism
Keywords: Dyspnea; Post-Pulmonary Embolism Syndrome
MeSH Terms: conditions — Dyspnea; Pulmonary Embolism | interventions — Nitric Oxide

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled crossover design
Who Masked: Participant, Investigator
Masking Description: Neither the participant, nor the clinical research coordinator conducting the exercise test will know which treatment is being administered. A separate, unblinded research associate will handle and administer treatment using the SoKINOX™ NO Delivery and Monitoring System
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Control (Placebo Comparator): Inhaled medical grade normoxic gas (FiO2 = 0.21; DIN 02238755 Air Liquid Healthcare, Montreal, Quebec, Canada).
  Interventions: Drug: Placebo
- Inhaled Nitric Oxide (Active Comparator): Inhaled 40 ppm nitric oxide from a KINOX™ gas cylinder system (Air Liquid Healthcare, Montreal, Quebec, Canada; Control # 198879, DIN 02451328).
  Interventions: Drug: Nitric Oxide

INTERVENTIONS:
Drug: Nitric Oxide — Pulmonary vasodilator (gas).
  Other Names: KINOX
  Arms: Inhaled Nitric Oxide
Drug: Placebo — medical grade normoxic gas (FiO2 = 0.21)
  Other Names: Medical Grade Air
  Arms: Placebo Control

SUMMARY:
Following acute pulmonary embolism (PE), up to a third of patients develop post-PE syndrome described as having persistent breathlessness (dyspnea), impaired exercise capacity, and a reduced quality of life. The post-PE syndrome includes patients with chronic thromboembolic pulmonary hypertension (CTEPH), patients with chronic thromboembolic disease (CTED) those with an obstruction of the pulmonary arteries without pulmonary hypertension, and patients with post-PE related dyspnea without obstruction or pulmonary hypertension. Although therapies exist for the most severe form of the post-PE syndrome (CTEPH) - for most patients there are no available disease specific therapies that reduce symptoms. Despite studies showing increased breathlessness and abnormal exercise responses in patients with CTED, a detailed examination of what causes breathlessness in post-PE syndrome has never been undertaken. It is suspected that reduced blood flow to the lungs contributes to the feelings of breathlessness, particularly during exercise.

This study will use inhaled nitric oxide, a medication that increases blood flow to the lungs. Inhaled nitric oxide is used primarily in hospitalized patients in the intensive care unit with respiratory failure, its use in people with post-PE syndrome is experimental. The investigators believe use of this medication may help to relieve symptoms of breathlessness. In order to test this medication, in volunteers with post-PE syndrome, the following will be measured: 1) breathlessness, 2) the signal to breathe sent from the brain to the lungs, 3) the activity of the muscles involved with breathing and 4) the amount of different gasses in the blood during exercise. The investigators will compare breathlessness and exercise tolerance during exercise while receiving: 1) a placebo (normal medical grade air) and 2) inhaled nitric oxide (a medication that improves blood flow to the lungs). By comparing symptoms during these two conditions, it is hoped to obtain a better understanding of what causes breathlessness in people with post-PE syndrome. This clinical research study will recruit approximately 20 clinically stable participants with CTED or post-PE related breathlessness.

DETAILED DESCRIPTION:
Background:

Following acute pulmonary embolism (PE), up to a third of patients develop post-PE syndrome characterized by persistent breathlessness (dyspnea), impaired exercise capacity, and reduced quality of life. Although therapies exist for the most severe manifestation of the post-PE syndrome [chronic thromboembolic pulmonary hypertension (CTEPH)] - for most patients there are no available disease specific therapies that reduce symptoms. In a preliminary study, it was observed that exertional dyspnea in post-PE syndrome was strongly associated with increased inspiratory neural drive (IND) to the diaphragm. High IND represents increased chemo-stimulation of medullary control centers due to the negative effects of increased ventilatory inefficiency measured as the ratio of ventilation to carbon-dioxide output (VE/VCO2). In a pilot study increased IND during exercise in the post-PE group was present despite the absence of measurable pulmonary hypertension at rest or exertional hypoxemia and was associated with increased VE/VCO2. The underlying mechanism for increased VE/VCO2 and IND during exercise in post-PE syndrome is currently unclear. Moreover, the contribution of adaptive changes by the respiratory controller, including altered chemosensitivity, to increased VE/VCO2 during exercise has not been determined. However, based on experiments to-date, the investigators propose that pulmonary microvascular abnormalities and hypoperfusion of pulmonary capillaries are potentially key pathophysiologic mechanisms. Accordingly, the purpose of the current application is to determine the degree of reversible vascular dysfunction that exists in these patients and to test the hypothesis that improved pulmonary gas exchange following an inhaled selective pulmonary vasodilator will reduce IND and exertional dyspnea intensity. The investigators plan to undertake a prospective, randomized, double-blind, placebo-controlled study of the effects of inhaled nitric oxide (iNO) on dyspnea intensity, IND, and physiologic responses to exercise to determine whether therapies acting on the NO pathway can reduce dyspnea and improve exercise capacity in the post-PE syndrome.

The post-PE syndrome encompasses the small minority of patients who develop CTEPH, defined as thrombotic occlusion of the pulmonary arteries with pulmonary hypertension. The post-PE syndrome also includes patients with chronic thromboembolic disease (CTED) with obstruction of the pulmonary arteries in the absence of pulmonary hypertension, and post-PE related dyspnea in patients with persistent symptoms in the absence of clear thrombotic occlusion or pulmonary hypertension.

Physiologic responses to exercise in the post-PE syndrome:

Cardiopulmonary exercise testing (CPET) is clinically useful in identifying CTEPH and deconditioning following PE. Exercise responses in CTEPH include increased ventilation (VE), dead space (regions of alveolar ventilation without perfusion), and VE/VCO2 as well as reduced peak oxygen uptake (VO2). Ventilatory inefficiency is increased in CTED and correlated with increased mean pulmonary artery pressure (mPAP)/cardiac output (CO) slope and physiological dead space.

Despite increased dyspnea and abnormal exercise responses, detailed neurophysiological mechanisms of dyspnea in the post-PE syndrome have not been undertaken. Accordingly, our recent study is the first to demonstrate that exertional dyspnea is increased in post-PE patients without resting pulmonary hypertension (Appendix I: Figure 1A) and highly correlated with magnitude of IND (r=0.761, p<0.01) (Figure 1B), secondary to elevated ventilatory demand during exercise (Figure 1C) in the absence of significant hypoxemia (Figure 1D). The current study extends our previous work by testing the strength of the association between high IND and high VE/VCO2 by selective pharmacological manipulation of the independent variable (VE/VCO2).

Extending CTEPH therapies to post-PE syndrome:

CTEPH is characterized by dual vascular abnormalities within the pulmonary artery tree: organized thromboembolic material in the large pulmonary arteries and a secondary vasculopathy in the small pulmonary arterioles with intimal thickening and remodeling. Surgical pulmonary endarterectomy (PEA) targets proximal pulmonary artery obstruction successfully in CTEPH with decrease in dead space, symptoms, and increased survival and has been extended to CTED. PEA however carries risk of complications occurring in up to 40% of patients perioperatively.

Multiple factors lead to small vessel vasculopathy in CTEPH including redirection of blood flow from areas obstructed by chronic emboli to non-obstructed vessels, contributing to pulmonary arteriole remodeling and altering endogenous NO production. Endogenous NO is synthesized by vascular endothelial cells, diffuses to vascular smooth muscle to activate soluble guanylate cyclase, and leads to smooth muscle relaxation. Medical treatment in inoperable or persistent CTEPH with Riociguat, a soluble guanylate cyclase stimulator, improves exercise capacity and reduces pulmonary vascular resistance (PVR) by acting in this pathway promoting smooth muscle relaxation. Due to rapid inactivation by heme moieties following administration, iNO acts in isolation on the pulmonary vasculature.

During right heart catheterization iNO is used in acute vasoreactivity testing for pulmonary hypertension. iNO decreases PVR and mPAP in animal models of acute pulmonary embolism and has been employed as adjunct therapy in intermediate risk acute PE in humans with improved residual volume (RV) function on echocardiography. Recent work has shown that iNO improved ventilatory efficiency (lower VE/VCO2) and exercise capacity (VO2peak) in mild chronic obstructive pulmonary disease (COPD) (manuscript in review). Although iNO in acute PE and the effect of vasodilators in CTEPH have been studied, to our knowledge manipulation of the physiologic responses to exercise in CTED and post-PE related dyspnea with iNO has not previously been undertaken.

Significance of the study:

The degree of pulmonary arteriole microvasculopathy and vascular dysfunction in the post-PE syndrome outside of CTEPH is an area of ongoing research. The common pattern of physiologic response to exercise in CTED and post-PE related dyspnea suggests that ventilatory inefficiency due to increased dead space plays a role in increased IND and exertional dyspnea throughout the spectrum of post-PE syndrome. Targeted manipulation of the pulmonary microvasculature to improve pulmonary blood flow and reduce dead space with iNO will allow for assessment of mechanisms of dyspnea and its relief in post-PE patients. A positive response to iNO will provide a physiological rationale for clinical assessment of medical therapies acting on the NO pathway in this population.

This proposed study will set the stage for new physiological studies to evaluate pulmonary vascular hemodynamics during exercise with echocardiography.

Trial Objectives:

Primary: To compare the acute effects of inhaled nitric oxide to placebo on dyspnea intensity (measured by 10-Point Borg Dyspnea Index) and inspiratory neural drive (IND) by diaphragm activation (EMGdi/EMGdi max) at rest, isotime and end-exercise during cardiopulmonary exercise testing (cycle ergometer).

Secondary: To compare the acute effects of inhaled nitric oxide to placebo on lung volumes, VE/VCO2 nadir, and dynamic respiratory mechanics at rest, isotime and end-exercise during cardiopulmonary exercise testing (cycle ergometer).

Hypothesis:

The following hypothesis will be tested 1) acute administration of inhaled nitric oxide (compared with placebo) will be associated with reduced VE/VCO2 nadir, IND, dyspnea, and increased exercise endurance time in patients with CTED or post-PE syndrome. The reduced ventilatory demand and breathing pattern alterations following inhaled vasodilator will be associated with delay in the onset of mechanical limitation to exercise.

ELIGIBILITY:
Inclusion Criteria:

1. clinically stable CTED or post-PE syndrome patients, as defined by stable hemodynamic status, optimized medical treatment, no changes in medication dosage or frequency of administration with no hospital admissions in the preceding 6 weeks;
2. a diagnosis of persistent, moderate to severe exertional dyspnea ≥ 6 months following PE as confirmed by study physician at time of enrollment by a modified Medical Research Council (mMRC) dyspnea scale =2, or Baseline Dyspnea Index (BDI) focal score <=6;
3. male or female non-pregnant adults >20 years of age;
4. ability to perform all study procedures
5. ability to provide informed consent

Exclusion Criteria:

1. women of childbearing potential who are pregnant or trying to become pregnant;
2. echocardiographic evidence of pulmonary hypertension
3. prior history of unstable pulmonary thromboembolism or systemic connective tissue vasculopathy,
4. active cardiopulmonary disease or other comorbidities that could contribute to dyspnea and exercise limitation;
5. history/clinical evidence of asthma, atopy and/or nasal polyps;
6. history of hypercapnic respiratory failure or a clinical diagnosis of sleep disordered breathing;
7. important contraindications to clinical exercise testing, including inability to exercise because of neuromuscular or musculoskeletal disease(s);
8. body mass index (BMI) <18.5 or ≥35.0 kg/m2;
9. use of daytime oxygen or exercise-induced O2 desaturation (<80% on room air).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Dyspnea Intensity | At isotime (maximum exercise time achieved by all participants during a standard CPET) from baseline (rest) up to 20 minutes.
  Dyspnea (respiratory discomfort) will be defined as the perceived "sensation of breathing discomfort" experienced at rest or during pedaling. Measurements will be made at rest (the steady-state period after at least 3 minutes of breathing on the mouthpiece before exercise starts), at two-minute intervals during exercise, and at end-exercise (at 2 minutes or the last 30-sec of loaded pedaling achieved by the participants). The intensity (strength) of sensations will be rated using the 10-point Borg scale (Modified Borg Dyspnoea Scale; scale from 0 to 10 in 1 unit increments, where 0 represents "Nothing at all" intensity and 10 represents "Maximal" intensity).
Leg discomfort Intensity | At isotime (maximum exercise time achieved by all participants during a standard CPET) from baseline (rest) up to 20 minutes..
  Leg discomfort will be defined as the perceived "sensation of leg discomfort" experienced at rest or during pedaling. Measurements will be made at rest (the steady-state period after at least 3 minutes of breathing on the mouthpiece before exercise starts), at two-minute intervals during exercise, and at end-exercise (at 2 minutes or the last 30-sec of loaded pedaling achieved by the participants). The intensity (strength) of sensations will be rated using the 10-point Borg scale (Modified Borg Dyspnoea Scale; scale from 0 to 10 in 1 unit increments, where 0 represents "Nothing at all" intensity and 10 represents "Maximal" intensity).
Inspiratory Neural Drive (IND) as measured by Diaphragmatic electromyography (EMGdi) | At isotime (maximum exercise time achieved by all participants during a standard CPET) from baseline (rest) up to 20 minutes..
  An esophageal electrode-balloon catheter consisting of 5 electrode pairs and two balloons, will be inserted nasally and positioned for optimal recording. Electromyogram output of the diaphragm (used as an index of inspiratory neural drive to crural diaphragm or diaphragm activation; EMGdi) will be recorded continuously at rest and during exercise. Maximal EMGdi (EMGdi,max) will be determined from IC maneuvers. EMGdi/EMGdi,max will be used as an index of the inspiratory neural drive to the crural diaphragm.

SECONDARY OUTCOMES:
Ventilation | At isotime (maximum exercise time achieved by all participants during a standard CPET) from baseline (rest) up to 20 minutes..
  Ventilation will be measured on a breath-by-breath basis using a SensorMedics Vmax229 metabolic measurement system. Measurements will be compared with predicted values based on age and height. Three main time points will be evaluated: "rest" defined as the steady-state period after at least 3 minutes of quiet breathing on the mouthpiece before exercise starts; "isotime" defined as the last 30-sec increment of each minute (i.e., 1-min, 2-min, 3-min) during the incremental exercise test and at 2 minutes (or the longest time achieved by all subjects) during the constant load exercise tests, and; "end-exercise" defined as the last 30-sec of loaded pedaling.
Respiratory Frequency | At isotime (maximum exercise time achieved by all participants during a standard CPET) from baseline (rest) up to 20 minutes..
  Respiratory frequency will be measured on a breath-by-breath basis using a SensorMedics Vmax229 metabolic measurement system. Measurements will be compared with predicted values based on age and height. Three main time points will be evaluated: "rest" defined as the steady-state period after at least 3 minutes of quiet breathing on the mouthpiece before exercise starts; "isotime" defined as the last 30-sec increment of each minute (i.e., 1-min, 2-min, 3-min) during the incremental exercise test and at 2 minutes (or the longest time achieved by all subjects) during the constant load exercise tests, and; "end-exercise" defined as the last 30-sec of loaded pedaling.
Inspiratory Capacity | At isotime (maximum exercise time achieved by all participants during a standard CPET) from baseline (rest) up to 20 minutes..
  Inspiratory capacity will be measured using a SensorMedics Vmax 229 metabolic measurement system. Measurements will be made at rest (the steady-state period after at least 3 minutes of breathing on the mouthpiece before exercise starts), at two-minute intervals during exercise, and at end-exercise (at 2 minutes or the last 30-sec of loaded pedaling achieved by the participants).
Carbon Dioxide Output (VECO2) | At isotime (maximum exercise time achieved by all participants during a standard CPET) from baseline (rest) up to 20 minutes..
  Carbon dioxide output (VECO2) will be measured on a breath-by-breath basis using a SensorMedics Vmax229 metabolic measurement system. Three main time points will be evaluated: "rest" defined as the steady-state period after at least 3 minutes of quiet breathing on the mouthpiece before exercise starts; "isotime" defined as the last 30-sec increment of each minute (i.e., 1-min, 2-min, 3-min) during the incremental exercise test and at 2 minutes (or the longest time achieved by all subjects) during the constant load exercise tests, and; "end-exercise" defined as the last 30-sec of loaded pedaling.
Oxygen Uptake (VEO2) | At isotime (maximum exercise time achieved by all participants during a standard CPET) from baseline (rest) up to 20 minutes..
  Oxygen uptake (VEO2) will be measured on a breath-by-breath basis using a SensorMedics Vmax229 metabolic measurement system. Three main time points will be evaluated: "rest" defined as the steady-state period after at least 3 minutes of quiet breathing on the mouthpiece before exercise starts; "isotime" defined as the last 30-sec increment of each minute (i.e., 1-min, 2-min, 3-min) during the incremental exercise test and at 2 minutes (or the longest time achieved by all subjects) during the constant load exercise tests, and; "end-exercise" defined as the last 30-sec of loaded pedaling.
Transdiaphragmatic pressure (Pdi) | At isotime (maximum exercise time achieved by all participants during a standard CPET) from baseline (rest) up to 20 minutes..
  An esophageal electrode-balloon catheter consisting of 5 electrode pairs and two balloons, will be inserted nasally and positioned for optimal recording. Esophageal (Pes) and gastric pressures (Pga) will be recorded continuously at rest and during exercise. Transdiaphragmatic pressure (Pdi) will be recorded as the difference between Pga and Pes signals.
Partial pressure of arterialized (capillary) carbon dioxide (PaCO2) | At isotime (maximum exercise time achieved by all participants during a standard CPET) from baseline (rest) up to 20 minutes..
  Earlobe arterialized blood will be collected at rest, and at end-exercise. Earlobe arterialized capillary blood gas sampling will be used to measure partial pressure of arterialized (capillary) carbon dioxide (PaCO2). PaCO2 values will be used to calculate ventilatory dead space.
Exercise Endurance Time | Time difference from start to isotime (maximum exercise time achieved by all participants) during a standard cardiopulmonary exercise test (cycle ergometer) up to 20 minutes.
  The time difference (in minutes and seconds) between the start of loaded pedaling until end-exercise (symptom limitation) of the cardiopulmonary exercise test performed on a stationary bicycle at 75% of maximum work rate.

CONTACTS AND LOCATIONS:
Overall Officials: Denis E O'Donnell, MD, Principal Investigator — Director Respiratory Investigation Unit, Professor
Locations (1):
- Respiratory Investigation Unit, Kingston General Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No